CLINICAL TRIAL: NCT06243393
Title: A Randomized, Open Label, Multicenter Phase II/III Trial of Sacituzumab Govitecan Compared to Standard of Care in Metastatic, Refractory Colorectal Cancer Patients
Brief Title: Sacituzumab Govitecan in Metastatic Colorectal Cancer
Acronym: TROPHIT1
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Bruno Christian Köhler, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT_GI_BCK_01; 2023-509771-17-00 (Other: EU CT Number); AIO-KRK-0124/ass (Other: AIO Germany)
Record Dates: First submitted 2024-01-24; First posted 2024-02-06 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan (SG) (Experimental): Treatment with Sacituzumab Govitecan (SG) .
  Interventions: Drug: Sacituzumab Govitecan (SG)
- Physicians Choice (PhC). (Active Comparator): Treatment according to oncologic guidelines.
  Interventions: Drug: Physicians Choice (PhC).

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Treatment with Sacituzumab Govitecan (SG)
  Arms: Sacituzumab Govitecan (SG)
Drug: Physicians Choice (PhC). — Treatment according to oncologic guidelines.
  Arms: Physicians Choice (PhC).

SUMMARY:
This is a Phase: II/III, open-label, multicenter (at least four centers in Germany) study of Sacituzumab Govitecan (SG) in metastatic colorectal cancer patients who are refractory to at least two lines of standard of care chemotherapy and not eligible for local therapy. There is no upper limit in the previous therapy lines. Patients must have documented progression or intolerability to combination chemotherapy including 5-fluoruacil or its prodrugs and derivates, Oxaliplatin and Irinotecan or a combination of the aforementioned. Previous biologicals/antibodies/small molecules including anti-EGFR and anti-VEGF directed therapies are allowed but not mandatory to meet eligibility. Trifluridin/Tipiracil (TAS102) or Regorafenib are allowed but not mandatory as previous therapies for PART I and PART II of the trial. All patients must have a documented Irinotecan-free interval of at least 6 months to be eligible for the study.

The study consists of two parts:

PART I: a single arm run in phase, treating 20 patients with Sacituzumab Govitecan (SG) PART II: a 1:1 randomized open label phase, comparing 30 patients treated with SG vs. 30 patients treated according to Physicians Choice (PhC). Crossover to the experimental arm (SG) is allowed in case of progression in the standard arm (PhC).

PART II will only be started if significant clinical efficacy and activity is observed in PART I.

ELIGIBILITY:
Inclusion Criteria

Patients meeting all of the following criteria are considered for admission to the trial:

1. Diagnosis of UICC Stage IV mCRC, not eligible for local therapy
2. Women or men aged ≥ 18 years, no upper age limit
3. ECOG performance status ≤2
4. Patients must have failed standard therapy or were intolerable towards standard therapy which must include fluoropyrimidine, oxaliplatin and irinotecan. (Targeted therapies (in combination with chemotherapy) including antiangiogenic monoclonal antibody/fusion protein/small molecule (e.g. bevacizumab, aflibercept, ramucirumab) and anti-EGFR antibody (e.g. Cetuximab, Panitumumab) are allowed as previous therapies.)
5. No Irinotecan treatment within the last 6 months. Patients that received Irinotecan treatment more than 6 months prior to inclusion, must have been responsive to Irinotecan induction therapy (i.e., patients previously exposed to induction chemotherapy containing irinotecan must have presented CR or PR or else SD at least 3 months or at initial response assessment).
6. At least one measurable lesion according to RECIST 1.1 that can be accurately assessed at screening by computed tomography or magnetic resonance imaging and is suitable for repeated assessment or available CT scan of thorax and abdomen not older than 30 days before start of treatment (day 1 of cycle 1).
7. Written informed consent
8. Non-pregnant and non-nursing women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to start of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile.

   Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   Post-menopausal or evidence of non-childbearing status is defined within this clinical trial:
   1. Amenorrhea for at least 12 consecutive months without an alternative medical cause following cessation of exogenous hormonal treatments.
   2. Chemotherapy-induced menopause with >1 year interval since last menses
   3. Surgical sterilisation
9. WOCBP are to be advised using two effective methods of birth control to avoid pregnancy throughout the study and for at least 6 months after the last dose of IMP. This includes effective contraception methods that can achieve a failure rate of less than 1% per year (e.g. hormonal contraceptive and condom, IUD/IUS and condom) or sterilization, resulting in a failure rate less than 1% per year.
10. Fertile men should not donate sperm and must be willing and able to use two effective methods of birth control (e.g latex condoms plus hormonal contraception in their partner) throughout the study and for at least 6 months after the last dose of IMP, if their sexual partners are WOCBP (acceptable methods see above). A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.

Exclusion Criteria

Patients meeting any of the following criteria are not eligible for the trial:

1. Patient with a known hypersensitivity to any of the excipients of sacituzumab govitecan
2. Participation in other clinical trials involving an investigational drug(s) (Phases 1-4) or observation period of competing trials, respectively within 4 weeks prior to study entry.

   Patients participating in observational studies are eligible.
3. Taking medications that may interfere with SN-38 metabolism.
4. Have had a prior anticancer biologic agent within 2 weeks prior to enrollment or have had prior chemotherapy, targeted therapy, or radiation therapy within 2 weeks prior to enrollment AND have not recovered (ie, ≥ Grade 2 is considered not recovered) from AEs at the time of study entry.
5. Have not recovered (ie, ≥ Grade 2 is considered not recovered) from AEs due to a previously administered agent.

   Note: patients with any grade neuropathy or alopecia are an exception to this criterion and will qualify for the study.

   Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Have an active second malignancy. Note: patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (eg, nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
7. History of significant cardiovascular disease ( NYHA ≥ III)
8. Clinical signs of active severe infection with or without requiring antibiotics.

   * Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load
   * Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.
   * Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
   * Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
9. Inadequate bone marrow, renal, and hepatic function defined by laboratory tests within 14 days prior to study treatment (growth factor support is not allowed within 14 days prior to baseline labs; Hemoglobin <9 g/dl, Neutrophil count <1500/ l, Platelet count <100000/l, Total bilirubin >1.5 times the institutional upper limit of normal (ULN, except patients with Gilbert Syndrome, there >3.0 mg/dl), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5 ULN; subjects with documented liver metastases may have an AST and ALT of >5.0 ULN and serum albumin <3 g/dl, Estimated creatinine clearance calculated creatinine clearance <30 ml/minute according to the Cockcroft and Gault formula)
10. Known microsatellite instable (MSI-H) / MMR-protein deficient (dMMR) colorectal cancer.
11. Any medical or other condition which, in the opinion of the Investigator, causes the subject to be medically unfit to receive sacituzumab govitecan, or unsuitable for any other reason
12. Pregnancy and lactation
13. Inability of patient to understand character and consequences of the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | time from randomization into the study to time of progression of the disease or death from any cause, whatever occurs first, assessed on average up to 1 year
  Progression Free Survival (PFS): as the time from randomization into the study to time of progression of the disease or death from any cause, whatever occurs first. Patients without an applicable event are censored on the last date of follow-up.

SECONDARY OUTCOMES:
Overall Survival (OS) | time from randomization into the study to time of death or end of study (EOS), assessed on average up to 1 year
  Overall Survival (OS): as time from randomization until death or end of study (EOS). Patients without an applicable event are censored on the last date of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided